CLINICAL TRIAL: NCT00003537
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Adult Patients With Anaplastic Astrocytoma
Brief Title: Antineoplaston Therapy in Treating Adult Patients With Anaplastic Astrocytoma
Acronym: AA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066585; BC-BT-8 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Adult Brain Tumor
Keywords: adult anaplastic astrocytoma
MeSH Terms: conditions — Brain Neoplasms; Astrocytoma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Adults with an anaplastic astrocytoma will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for adults with anaplastic astrocytoma provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of adults with anaplastic astrocytoma.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on adults with anaplastic astrocytoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in adults with anaplastic astrocytoma as measured by an objective response to therapy (complete response, partial response) or stable disease.
* To determine the safety and tolerance of Antineoplaston therapy in adults with anaplastic astrocytoma.

OVERVIEW: This is a single arm, open-label study in which adults with anaplastic astrocytoma receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with a complete or partial response or with stable disease may continue treatment.

To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of anaplastic astrocytoma
* Tumor subtotally resected or biopsied prior to therapy
* Evidence of residual tumor by MRI scan performed within two weeks prior to study entry
* No brain stem tumors

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 2 months

Hematopoietic:

* WBC at least 1,500/mm^3
* Platelet count at least 50,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No renal failure

Cardiovascular:

* No prior congestive heart failure
* No coronary artery disease
* No myocardial infarction within the past year
* No angina requiring medication
* No uncontrolled hypertension

Pulmonary:

* No moderate to severe chronic obstructive pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No active infection
* No other concurrent serious disease
* No other prior malignancy except carcinoma in situ of the cervix or superficial nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy
* No concurrent immunomodulating agents

Chemotherapy:

* No prior myelosuppressive chemotherapy

Endocrine therapy:

* Concurrent corticosteroids for cerebral edema allowed

Radiotherapy:

* No prior myelosuppressive radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from any prior surgery

Other:

* No prior cytodifferentiating agents
* No prior antineoplaston therapy
* No other concurrent antineoplastic agents

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1995-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burzynski SR, Janicki TJ, Burzynski GS, Marszalek A. A Phase II Study of Antineoplastons A10 and AS2-1 in Adult Patients with Newly-Diagnosed Anaplastic Astrocytoma Final Report (Protocol BT-08). Cancer and Clinical Oncology 4: 28-38, 2015. DOI: http://dx.doi.org/10.5539/cco.v4n1p28
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nineteen patients were recruited between April 1995 and October 2008. All study subjects were seen at the Burzynski Clinic in Houston TX
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Adults with a residual or recurrent anaplastic astrocytoma will receive Antineoplaston therapy (Atengenal + Astugenal).
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 19
Completed | 18
Not Completed | 1
Not completed — Not evalauable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: Years] | 44.0 [22.4 to 60.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks; Stable Disease (SD), <50% decrease and <25% increase in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least eight weeks; Progressive Disease (PD), >=25% increase in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 18
Participants
  Complete Response | 3
  Partial Response | 1
  Stable Disease | 5
  Progressive Disease | 9

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 19
Percentage of participants
  6 months overall survival | 68.4
  12 months overall survival | 52.6
  24 months overall survival | 36.8
  36 months overall survival | 26.3
  48 months overall survival | 26.3
  60 months overall survival | 21.1

ADVERSE EVENTS:
Time Frame: 13 years, 6 months
Description: Nineteen patients were recruited between April 1995 and October 2008. All study subjects were seen at the Burzynski Clinic in Houston TX
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 11/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=19)
Supraventricular and nodal arrhythmia: Atrial fibrillation (Cardiac disorders) | 1 — The Supraventricular and nodal arrhythmia: Atrial fibrillation was not related to Antineoplaston therapy.
Ventricular arrhythmia: Ventricular tachycardia (Cardiac disorders) | 1 — The Ventricular arrhythmia: Ventricular tachycardia was not related to Antineoplaston therapy.
Hypotension (Cardiac disorders) | 1 — Th hypotension was not related to Antineoplaston therapy.
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 — The Pericardial effusion (non-malignant) was not related to Antineoplaston therapy.
Central venous catheter infection (General disorders) | 4 — The Central venous catheter infections were not related to Antineoplaston therapy
Thrombosis/embolism (General disorders) | 1 — The Thrombosis/embolism was not related to Antineoplaton therapy.
Fever (General disorders) | 2 — The Fevers were not related to Antineoplaston therapy.
Rigors/chills (General disorders) | 2 — The Rigors/chills were not related to Antineoplaston therapy.
Hemorrhage, CNS (Nervous system disorders) | 1 — The Hemorrhage, CNS was not related to Antineoplaston therapy.
Infection (documented clinically): Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 3 — The Infections (documented clinically): Lung (pneumonia) were not related to Antineoplaston therapy.
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 1 — The Infection (documented clinically): Bladder (urinary) was not related to Antineoplaston therapy.
Hypokalemia (Investigations) | 1 — The Hypokalemia was not related to Antineoplaston therapy.
Neuropathy: motor (Nervous system disorders) | 1 — The Neuropathy: motor was not related to Antineoplaston therapy.
Seizure (Nervous system disorders) | 2 — The Seizures were not related to Antineoplaston therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 3 — The Somnolences/depressed levels of consciousness were not related to Antineoplaston therapy.
Diplopia (Eye disorders) | 1 — The diplopia was not related to Antineoplaston therapy.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 — The Pneumothorax was not related to Antineoplaston therapy.
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 — The Thrombosis/embolism (vascular access-related) was not related to Antineoplaston therapy.
Thrombosis/thrombus/embolism (Vascular disorders) | 1 — The Thrombosis/thrombus/embolism was not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=19)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 6
Auditory/Ear - Other (Ear and labyrinth disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 5
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 7
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2
Platelets (Blood and lymphatic system disorders) | 3
Palpitations (Cardiac disorders) | 2
Supraventricular and nodal arrhythmia: Atrial fibrillation (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia: Sinus tachycardia (Cardiac disorders) | 1
Ventricular arrhythmia: Ventricular tachycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 3
Hypotension (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 1
Central venous catheter infection (Infections and infestations) | 6
Non-functional central venous catheter (General disorders) | 6
Central venous catheter - Other (General disorders) | 6
Pain: Central venous catheter (General disorders) | 2
Central venous catheter thrombosis/embolism (General disorders) | 5
Fatigue (asthenia, lethargy, malaise) (Gastrointestinal disorders) | 9
Fever (General disorders) | 5
Rigors/chills (General disorders) | 4
Sweating (diaphoresis) (General disorders) | 1
Weight gain (General disorders) | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Edema/Fluid retention (General disorders) | 8
Diarrhea (Gastrointestinal disorders) | 4
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 7
Hemorrhage, CNS (Nervous system disorders) | 1
Hemorrhage, GU: Bladder (Renal and urinary disorders) | 1
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Infection - Other (Infections and infestations) | 1
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 4
Infection (documented clinically): Middle ear (otitis (Infections and infestations) | 1
Infection (documented clinically): Blood (Infections and infestations) | 1
Infection (documented clinically): Bronchus (Infections and infestations) | 1
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 4
Infection (documented clinically): Mucosa (Infections and infestations) | 3
Infection (documented clinically): Neck NOS (Infections and infestations) | 1
Infection (documented clinically): Oral cavity-gums (gingivitis) (Infections and infestations) | 1
Infection (documented clinically): Sinus (Infections and infestations) | 1
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 3
Opportunistic infection (Infections and infestations) | 1
Edema:head and neck (Blood and lymphatic system disorders) | 1
Albumin, serum-low (hypoalbuminemia) (Investigations) | 2
Alkaline phosphatase (Investigations) | 3
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 3
Hyperbilirubinemia (Investigations) | 1
Hypercalcemia (Investigations) | 2
Hypercholesteremia (Investigations) | 2
Hyperglycemia (Investigations) | 7
Hypernatremia (Investigations) | 12
Hypertriglyceridemia (Investigations) | 3
Hyperuricemia (Investigations) | 1
Hypocalcemia (Investigations) | 4
Hypokalemia (Investigations) | 18
Hypoglycemia (Investigations) | 5
Hypomagnesemia (Investigations) | 1
Hyponatremia (Investigations) | 1
Hypophosphatemia (Investigations) | 4
Metabolic/Laboratory - Other (Investigations) | 1
Proteinuria (Renal and urinary disorders) | 5
SGOT (Investigations) | 7
SGPT (Investigations) | 8
Uric acid, serum-high (hyperuricemia) (Investigations) | 1
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1
Ataxia (incoordination) (Nervous system disorders) | 2
Confusion (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 3
Mood alteration (Nervous system disorders) | 2
Mood alteration: Agitation (Nervous system disorders) | 2
Neurology - Other (Nervous system disorders) | 1
Mood alteration: Anxiety (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 4
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1
Pyramidal tract dysfunction (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 6
Somnolence/depressed level of consciousness (Nervous system disorders) | 10
Speech impairment (Nervous system disorders) | 4
Diplopia (Ear and labyrinth disorders) | 2
Nystagmus (Eye disorders) | 2
Vision-blurred vision (Eye disorders) | 5
Vision-photophobia (Eye disorders) | 1
Pain: Abdomen NOS (Gastrointestinal disorders) | 1
Pain: Back (Musculoskeletal and connective tissue disorders) | 2
Pain: Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1
Pain: External ear (Ear and labyrinth disorders) | 1
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain: Head/headache (Nervous system disorders) | 13
Pain: Joint (Musculoskeletal and connective tissue disorders) | 6
Pain: Middle ear (Ear and labyrinth disorders) | 1
Pain: Muscle (Metabolism and nutrition disorders) | 2
Pain: Neck (Musculoskeletal and connective tissue disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 5
Flu-like syndrome (Infections and infestations) | 3
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 2
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No